CLINICAL TRIAL: NCT00911443
Title: A Phase II, Multicentre, Open, Randomised, Dose Ranging Study to Investigate the Efficacy of Combination Therapy Containing Dacarbazine (DTIC) Plus Low Dose Interferon Alpha (aIFN) Plus Thymosin a1 Versus Both DTIC Plus Thymosin a1 and DTIC Plus aIFN in Patients With Advanced -Stage Metastatic Malignant Melanoma
Brief Title: Thymosin Alpha 1, Interferon Alpha, or Both, in Combination With Dacarbazine in Patients With Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: sigma-tau i.f.r. S.p.A. (Industry)
Responsible Party: ROBERTO CAMERINI / Head of Clinical Research II, sigma-tau i.f.r. S.p.A.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST1472DM01012
Record Dates: First submitted 2009-02-26; First posted 2009-06-02 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Dacarbazine; Interferon-alpha; Thymalfasin; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dacarbazine + Interferon alpha + thymosin-alpha-1 1.6 mg (Experimental): Dacarbazine 800 mg/m2 IV on day 1; Interferon alpha 3MIU SC on day 11 and 18; Thymosin-alpha-1 1.6 mg SC from day 8 to 11 and from day 15 to 18 of each 28 day cycle up to 6 cycles or until progression or unacceptable toxicity develops.
  Interventions: Biological: Dacarbazine + Interferon alpha + Thymosin-alpha-1 1.6 mg
- Dacarbazine + Interferon alpha + Thymosin-alpha-1 3.2 mg (Experimental): Dacarbazine 800 mg/m2 IV on day 1; Interferon alpha 3MIU SC on day 11 and 18; Thymosin-alpha-1 3.2 mg SC from day 8 to 11 and from day 15 to 18 of each 28 day cycle up to 6 cycles or until progression or unacceptable toxicity develops.
  Interventions: Biological: Dacarbazine + Interferon alpha + Thymosin-alpha-1 3.2 mg
- Dacarbazine + Interferon alpha + Thymosin-alpha-1 6.4 mg (Experimental): Dacarbazine 800 mg/m2 IV on day 1; Interferon alpha 3MIU SC on day 11 and 18; Thymosin-alpha-1 6.4 mg SC from day 8 to 11 and from day 15 to 18 of each 28 day cycle up to 6 cycles or until progression or unacceptable toxicity develops.
  Interventions: Biological: Dacarbazine + Interferon alpha + Thymosin-alpha-1 6.4 mg
- Dacarbazine + Thymosin-alpha-1 3.2 mg (Experimental): Dacarbazine 800 mg/m2 IV on day 1; Thymosin-alpha-1 3.2 mg SC from day 8 to 11 and from day 15 to 18 of each 28 day cycle up to 6 cycles or until progression or unacceptable toxicity develops.
  Interventions: Biological: Dacarbazine + Thymosin-alpha-1 3.2 mg
- Dacarbazine + Interferon alpha (Active Comparator): Dacarbazine 800 mg/m2 IV on day 1; Interferon alpha 3MIU SC on day 11 and 18 of each 28 day cycle up to 6 cycles or until progression or unacceptable toxicity develops.
  Interventions: Drug: Dacarbazine + Interferon alpha

INTERVENTIONS:
Biological: Dacarbazine + Interferon alpha + Thymosin-alpha-1 1.6 mg — Dacarbazine 800 mg/m2 IV on day 1;Interferon alpha 3MIU SC on day 11 and 18; Thymosin-alpha-1 1.6 mg SC from day 8 to 11 and from day 15 to 18 of each 28 day cycle up to 6 cycles or until progression or unacceptable toxicity develops.
  Other Names: Zadaxin; Thymalfasin; ST1472; Deticene; Roferon
  Arms: Dacarbazine + Interferon alpha + thymosin-alpha-1 1.6 mg
Biological: Dacarbazine + Interferon alpha + Thymosin-alpha-1 3.2 mg — Dacarbazine 800 mg/m2 IV on day 1; Interferon alpha 3MIU SC on day 11 and 18; Thymosin-alpha-1 3.2 mg SC from day 8 to 11 and from day 15 to 18 of each 28 day cycle up to 6 cycles or until progression or unacceptable toxicity develops.
  Other Names: Zadaxin; Thymalfasin; ST1472; Deticene; Roferon
  Arms: Dacarbazine + Interferon alpha + Thymosin-alpha-1 3.2 mg
Biological: Dacarbazine + Interferon alpha + Thymosin-alpha-1 6.4 mg — Dacarbazine 800 mg/m2 IV on day 1; Interferon alpha 3MIU SC on day 11 and 18 Thymosin-alpha-1 6.4 mg SC from day 8 to 11 and from day 15 to 18 of each 28 day cycle up to 6 cycles or until progression or unacceptable toxicity develops.
  Other Names: Zadaxin; Thymalfasin; ST1472; Deticene; Roferon
  Arms: Dacarbazine + Interferon alpha + Thymosin-alpha-1 6.4 mg
Biological: Dacarbazine + Thymosin-alpha-1 3.2 mg — Dacarbazine 800 mg/m2 IV on day 1; Thymosin-alpha-1 3.2 mg SC from day 8 to 11 and from day 15 to 18 of each 28 day cycle up to 6 cycles or until progression or unacceptable toxicity develops.
  Other Names: Zadaxin; Thymalfasin; ST1472; Deticene
  Arms: Dacarbazine + Thymosin-alpha-1 3.2 mg
Drug: Dacarbazine + Interferon alpha — Dacarbazine 800 mg/m2 IV on day 1; Interferon alpha 3MIU SC on day 11 and 18 of each 28 day cycle up to 6 cycles or until progression or unacceptable toxicity develops.
  Other Names: Deticene; Roferon
  Arms: Dacarbazine + Interferon alpha

SUMMARY:
The purpose of the study is to test safety and efficacy of different doses of thymosin alpha 1 (1.6 mg, 3.2 mg, and 6.4 mg) in combination with dacarbazine and with or without Interferon alpha in treating patients affected by stage IV melanoma.

Primary end-point is Tumor Response evaluated according to Response Evaluation Criteria In Solid Tumors (RECIST). Secondary end-points are Overall Survival and Progression Free Survival.

Ninety-five patients are allocated to each arm to test the hypothesis that P0 <= 0.05 vs the alternative hypothesis that P1 >= 0.15 (alpha = 5%, within-group statistical analysis beta = 95%).

ELIGIBILITY:
Inclusion Criteria:

* Have read and signed the informed consent form
* 18 years <=Age<= 75 years
* Adequate contraception practice (fertile female patient)
* Confirmed diagnosis of metastatic melanoma (stage IV) with unresectable metastases and >= 1 measurable lesion
* Adequate renal function as demonstrated by serum creatinine level < 1.5 mg/deciliter (dl)
* Absolute Neutrophil Count (ANC) >= 1.5 x 10000000000/L ; platelets >= 100 x 10000000000/Liter (L)
* Good performance status: PS <= 1 (ZUBROD-ECOG-WHO scale)
* At least 12 week life expectancy

Exclusion Criteria:

* Clinical diagnosis of autoimmune disease
* Transplant recipient
* Pregnancy documented by a urine pregnancy test or lactation
* Previous treatment with thymosin alpha 1
* Previous treatment with chemotherapy
* Presence of Central Nervous System (CNS) metastases
* Concomitant or prior history of malignancy other than melanoma
* Participation in another investigational trial within 30 days of study entry
* Active infectious process that is not of self-limiting nature

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2002-07; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Ferraresi, MD, Principal Investigator — IFO Polo Oncologico Ist. Regina Elena, Divisione Oncologia Medica A - ROMA; Roberto Camerini, MD, Study Director — Sigma-Tau SpA
Locations (64):
- France (5):
  - CHU de Grenoble Hopital Albert Michallon Service de Dermatologie, La Tronche
  - CHU de Limoges Hopital Dupuytren Service de Dermatologie, Limoges
  - Hopital Saint-Eloi Service de Dermatologie, Montpellier
  - Centre Eugene Marquis Departement d'Oncologie Medicale, Rennes
  - Hopital Purpan Service de Dermatologie, Toulouse
- Germany (8):
  - Klinik fur Dermatologie und Allergologie der RWTH Aachen, Aachen
  - Klinik fur Dermatologie, Venerologie und Allergologie des Campus Charitè Mitte, Berlin
  - Elbeklinikec Buxtehude Dermatologische Zentrum Abteilung fur Dermato-Onkologie, Buxtehude
  - Zentrum fur Dermatologie und Veneralogie Klinik der Johann-Wolfgang-Goethe-Universitat, Frankfurt
  - Klinikum Hannover, Hautklinik Linden, Hanover
  - Universitatsklinikum Schlewig-Holstein Klinik fur Dermatologie, Veneralogie und Allergologie Universitats-Hautklinik Kiel, Kiel
  - Universitatsklinik fur Dermatologie und Venerologie Otto-von-Guericke-Universitat Magdeburg, Magdeburg
  - Dermatologische Klinik der Universitat Tubingen, Tübingen
- Hungary (6):
  - Orszagos Bor-es Nemikortani Intezet, Budapest
  - Orszagos Onkologiai Intezet Borgyogyaszat, Budapest
  - Petz Aladar Megyei Korhaz, Borgyogyaszat, Győr
  - Miskolc Megyei Korhaz Borgyogyaszat, Miskolc
  - Pecsi Egyetem Borgyogyaszati Klinika, Pécs
  - Szegedi Egyetem Borgyogyaszati Klinika, Szeged
- Italy (25):
  - Ospedale SS Trinità Oncologia, Sora, FROSINONE
  - Ospedale San Vincenzo U.O. Oncologia Medica, Taormina, MESSINA
  - UO Complessa Aziendale Nettuno/Albano/Frascati Day-Hospital di Oncologia Ospedale S. Giuseppe, Albano Laziale, ROMA
  - Ospedale PF Calvi Dipartimento di Oncologia, Noale, VENEZIA
  - ASL 1 Servizio di Oncologia, Agrigento
  - Azienda Ospedaliera S. Elia, UO di Oncologia, Caltanissetta
  - Azienda Ospedaliera Garibaldi, UO Oncologia Medica, Catania
  - Università "G. D'Annunzio" Facoltà di Medicina e Chirurgia, Clinica Dermatologica, Chieti
  - Azienda Ospedaliera Umberto I° UO Servizio di Oncologia e Chemioterapia, Enna
  - Università di Firenze Dipartimento di Scienze Dermatologiche, Florence
  - Ospedale Pierantoni, Divisione Oncologia Medica, Forlì
  - Istituto NazionaleRicerca sul Cancro, Dipartimento di Oncologia Medica 1, Genova
  - Istituto Europeo di Oncologia, Divisione di Chirurgia Generale, Milan
  - Casa di Cura San Pio X, UO Oncologia Medica, Milan
  - Ospedale Civile, UO di Oncologia, Ragusa
  - Azienda Ospedaliera Bianchi-Melacrino-Morelli, Oncologia Medica, Reggio Calabria
  - Università di Roma "Tor Vergata" Oncologia Complementare, Dipartimento di Chirurgia, Roma
  - IFO Polo Oncologico Ist. Regina Elena, Divisione di Oncologia Medica A, Roma
  - Ospedale Sandro Pertini, Oncologia Medica, Roma
  - Università "La Sapienza" Dipartimento di Malattie Cutanee-Veneree e Chirurgia Plastica Ricostruttiva, Roma
  - Istituto Dermopatico dell'Immacolata, Dipartimento di Immunodermatologia, Roma
  - Policlinico "Le Scotte" Dipartimento di Medicina Clinica, Scienze Immunologiche Applicate, Divisione di Dermatologia, Siena
  - U.O. Complessa, Immunoterapia Oncologica, Policlinico "Le Scotte", Siena
  - Ospedale Umberto I°, Divisione di Oncologia Medica, Syracuse
  - Ospedale Bel Colle UO di Oncologia, Viterbo
- Poland (8):
  - Katedra i Klinika Onkologii i Radioterapii Akademia Medyczna, Gdansk
  - Instytut Onkologii im. Marii Sklodowskiej-Curie, Oddzial w Krakowie, Klinika Chemioterapii, Krakow
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika, Klinika Chemioterapii Oncologicznej, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 1, Klinika Chirurgii Onkologicznej, Lublin
  - Wielkopolskie Centrum Onkologii, Zaklad Immunologii Nowotworow Katedry Onkologii AM, Poznan
  - Oddzial Chemioterapii, Szczecin
  - Klinika Onkologii Centralnego Szpitala WAM, Warsaw
  - Dolnoslakie Centrum Transplantacji Komorkowych z Krajowym Bankiem Dawcow Szpiku, Wroclaw
- Portugal (2):
  - Instituto Portugues de Oncologia de Francisco Gentil, Centro Regional de Oncologia de Lisboa S.A., Servicio de Medicina Oncologica 1, Pavilhao C, Lisbon
  - Instituto Portugues de Oncologia de Francisco Gentil, Centro Regional de Oncologia do Porto S.A., Servicio de Medicina Oncologica, Piso 3, Porto
- Spain (9):
  - Instituto Catalan Oncologico, Servicio de Oncologia, L'Hospitalet de Llobregat, BARCELONA
  - Hosp. Univ. de Canarias Servicio de Oncologia Medica, San Cristóbal de La Laguna, SANTA CRUZ DE TENERIFE
  - Hosp. Clinic i Provincial Servicio de Oncologia, Barcelona
  - Hosp. Universitario de Jaen Servicio de Oncologia, Jaén
  - Hosp. Clinico San Carlos Servicio de Oncologia, Pabellon B, Ala Sur-Sotano, Madrid
  - Hosp. Virgen de la Victoria de Malaga Servicio de Oncologia 1a planta Campus Universitario de Teatinos, Málaga
  - Hosp. Virgen del Rocio Servicio de Oncologia, Planta Baja - Centro de Diagnostico, Seville
  - Instituto Valenciano Oncologico, Valencia
  - Hospital General Universitario de Valencia Unidad de Oncologia Medica, Valencia
- Zentrum fur Onkologie Hematologie und Transfusionsmedizin am Kantonsspital Aarau, Aarau, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on August 2002 and has been completed on January 2006. All patients were recruited at medical clinic facilities (Oncology/Dermatology departments)
Pre-assignment Details: Only patients who did not meet the entry selection criteria were excluded from study entry.
Groups:
- Dacarbazin + Interferon Alpha + Thymosin-alpha-1 1.6 mg: Dacarbazin 800 mg/m2 IV on day 1; Interferon alpha 3MIU SC on day 11 and 18; Thymosin-alpha-1 1.6 mg SC from day 8 to 11 and from day 15 to 18 of each 28 day cycle up to 6 cycles or until progression or unacceptable toxicity develops.
- Dacarbazin + Interferon Alpha + Thymosin-alpha-1 3.2 mg: Dacarbazin 800 mg/m2 IV on day 1; Interferon alpha 3MIU SC on day 11 and 18; Thymosin-alpha-1 3.2 mg SC from day 8 to 11 and from day 15 to 18 of each 28 day cycle up to 6 cycles or until progression or unacceptable toxicity develops.
- Dacarbazin + Interferon Alpha + Thymosin-alpha-1 6.4 mg: Dacarbazin 800 mg/m2 IV on day 1; Interferon alpha 3MIU SC on day 11 and 18; Thymosin-alpha-1 6.4 mg SC from day 8 to 11 and from day 15 to 18 of each 28 cycle up to 6 cycles or until progression or unacceptable toxicity develops.
- Dacarbazin + Thymosin-alpha-1 3.2 mg: Dacarbazin 800 mg/m2 IV on day 1; Thymosin-alpha-1 3.2 mg SC from day 8 to 11 and from day 15 to 18 of each 28 day cycle up to 6 cycles or until progression or unacceptable toxicity develops.
- Dacarbazin + Interferon Alpha: Dacarbazin 800 mg/m2 IV on day 1; Interferon alpha 3MIU SC on day 11 and 18 of each 28 day cycle up to 6 cycles or until progression or unacceptable toxicity develops.
Period: Overall Study
Arm/Group | Dacarbazin + Interferon Alpha + Thymosin-alpha-1 1.6 mg | Dacarbazin + Interferon Alpha + Thymosin-alpha-1 3.2 mg | Dacarbazin + Interferon Alpha + Thymosin-alpha-1 6.4 mg | Dacarbazin + Thymosin-alpha-1 3.2 mg | Dacarbazin + Interferon Alpha
Started | 97 | 97 | 98 | 99 | 97
Completed | 97 | 97 | 98 | 99 | 97
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dacarbazin + Interferon Alpha + Thymosin-alpha-1 1.6 mg | Dacarbazin + Interferon Alpha + Thymosin-alpha-1 3.2 mg | Dacarbazin + Interferon Alpha + Thymosin-alpha-1 6.4 mg | Dacarbazin + Thymosin-alpha-1 3.2 mg | Dacarbazin + Interferon Alpha | Total
Number analyzed (Participants) | 97 | 97 | 98 | 99 | 97 | 488
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0.0
  Between 18 and 65 years | 69 | 69 | 67 | 73 | 68 | 346.0
  >=65 years | 28 | 28 | 31 | 26 | 29 | 142.0
Age Continuous [Mean (Standard Deviation); unit: years] | 54 (14) | 54 (14) | 56 (13) | 56 (11) | 57 (12) | 55 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 50 | 45 | 38 | 55 | 226.0
  Male | 59 | 47 | 53 | 61 | 42 | 262.0
Region of Enrollment [Number; unit: participants]
  France | 14 | 7 | 11 | 6 | 5 | 43.0
  Portugal | 0 | 0 | 0 | 0 | 1 | 1.0
  Hungary | 3 | 4 | 1 | 2 | 9 | 19.0
  Spain | 4 | 2 | 2 | 13 | 6 | 27.0
  Poland | 26 | 28 | 32 | 36 | 37 | 159.0
  Germany | 17 | 22 | 25 | 10 | 11 | 85.0
  Switzerland | 0 | 0 | 0 | 1 | 0 | 1.0
  Italy | 33 | 34 | 27 | 31 | 28 | 153.0

OUTCOME MEASURES:

1. Secondary Outcome: Overall Survival
Description: The survival time for each patient is defined as the time between randomization and death. Patients lost to follow-up or still alive at the date of last evaluation have been censored.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacarbazin + Interferon Alpha + Thymosin-alpha-1 1.6 mg | Dacarbazin + Interferon Alpha + Thymosin-alpha-1 3.2 mg | Dacarbazin + Interferon Alpha + Thymosin-alpha-1 6.4 mg | Dacarbazin + Thymosin-alpha-1 3.2 mg | Dacarbazin + Interferon Alpha
Number analyzed (Participants) | 97 | 97 | 98 | 99 | 97
months | 9.3 [8.0 to 11.1] | 8.6 [6.1 to 11.6] | 10.3 [8.2 to 12.7] | 9.3 [6.7 to 11.7] | 6.6 [5.3 to 9.9]

2. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival is defined as the time from the randomization to progression or death
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacarbazin + Interferon Alpha + Thymosin-alpha-1 1.6 mg | Dacarbazin + Interferon Alpha + Thymosin-alpha-1 3.2 mg | Dacarbazin + Interferon Alpha + Thymosin-alpha-1 6.4 mg | Dacarbazin + Thymosin-alpha-1 3.2 mg | Dacarbazin + Interferon Alpha
Number analyzed (Participants) | 97 | 97 | 98 | 99 | 97
months | 1.9 [1.8 to 2.6] | 1.8 [1.8 to 2.0] | 1.8 [1.8 to 2.6] | 2.0 [1.8 to 3.5] | 1.8 [1.7 to 2.0]

3. Primary Outcome: Overall Tumor Response
Description: Tumor response is measured according to Response Evaluation Criteria In Solid Tumors (RECIST) computing number of Complete Response plus Partial Response
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Dacarbazin + Interferon Alpha + Thymosin-alpha-1 1.6 mg | Dacarbazin + Interferon Alpha + Thymosin-alpha-1 3.2 mg | Dacarbazin + Interferon Alpha + Thymosin-alpha-1 6.4 mg | Dacarbazin + Thymosin-alpha-1 3.2 mg | Dacarbazin + Interferon Alpha
Number analyzed (Participants) | 97 | 97 | 98 | 99 | 97
participants | 7 | 10 | 6 | 12 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less